CLINICAL TRIAL: NCT02950727
Title: Stability of Bilateral Sagittal Split Ramus Osteotomy (BSSRO) Using Adjustable Mandibular Plates in Adjunction With Bicortical Screws Versus Traditional Positional Screws for Antero-posterior Mandibular Deficient Patients
Brief Title: Comparing Stability and Cost-Effectiveness of 3 Bicortical Screws Vs Adjustable Plate and 2 Bicortical Screws in Fixation of BSSRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph Van Sickels (Other)
Responsible Party: Sponsor-Investigator, Joseph Van Sickels, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-0769-F3R
Record Dates: First submitted 2016-08-23; First posted 2016-11-01 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Mandibular Hypoplasia
Keywords: orthognathic surgery; bicortical screws; monocortical plates
MeSH Terms: conditions — Micrognathism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 bicortical screw (Experimental): 1st group:3 bicortical screws will be used to fix the sagittal split ramus osteotomy.
  Interventions: Device: 3 bicortical screws
- adjustable plate and 2 bicortical screws (Active Comparator): adjustable plate and 2 bicortical screws will be used to fix the sagittal split ramus osteotomy.
  Interventions: Device: adjustable plate and 2 bicortical screws

INTERVENTIONS:
Device: 3 bicortical screws — after mandibular bilateral sagittal split ramus osteotomy surgery is performed in the first group the osteotomy will be fixed using 3 bicortical screws
  Arms: 3 bicortical screw
Device: adjustable plate and 2 bicortical screws — after mandibular bilateral sagittal split ramus osteotomy surgery is performed in the second group the osteotomy will be fixed using adjustable plate and 2 bicortical screws
  Arms: adjustable plate and 2 bicortical screws

SUMMARY:
In this current study a comparison between 3 positional screws versus the adjustable plating system in conjunction with 2 positional screws. The patients will be selected to have retrognathic mandible requiring advancement. Hypothetically the advantage of the adjustable plating system will be compared with the three positional screws. In theory, the investigators will be using the inherent advantage of the intraoperative flexibility of the adjustable plating system in verifying the position of the proximal segment (condylar segment), hence eliminating the immediate postoperative relapse that is reported with using three positional screws. This will be evaluated both clinically and cephalometrically.

DETAILED DESCRIPTION:
Trauner and Obwegeser in 1957, reported the first correction of jaw deformity by the sagittal split technique.

Dal Pont in 1961, a student of Obwegeser, made a modification to the latter technique, to further enhance the precision and the accuracy of movement of both proximal distal segments his technique has become widely publicized. He changed the lower horizontal cut to a vertical cut on the buccal cortex between the first and second molars, there by obtaining broader bony contact.

Hunsuck in 1968, modified the technique, to decrease the soft tissue dissection; he advocated a shorter horizontal medial cut.

Epker in 1977, modified the technique in several ways to decrease swelling, manipulation to the neurovascular bundle and hemorrhage, his modification included minimal stripping of the masseter muscle and medial dissection.

BSSRO is now the most common procedure used to advance the mandible is a bilateral sagittal split osteotomy.

There are many different methods of mandibular fixation such as using intra osseous wiring combined with inter maxillary fixation (IMF) which showed significant amount of relapse and patient dissatisfaction, this is called nonrigid fixation. Another type of mandibular fixation is the three point fixation using positioning screws called rigid fixation. Rigid internal fixation was introduced in 1976 by Spiessel to promote healing, restore early function, and decrease relapse. The introduction of an internal rigid fixation method, instead of 5-6 week intermaxillary fixation, had the added benefit of shorter periods of hospital stay and patient convenience.' Minimal or no immobilization of the jaws allows patients to function sooner, resume their daily activities, and return to work earlier. In a relatively short period of time, the use of rigid fixation of bony segments in orthognathic surgery had become a standard of care.

A major concern in the surgical correction of a anteroposterior mandibular deficient patients is potential postsurgical relapse.

Clinical studies have shown a wide array of successful techniques used to fix segments. Three bicortical screws placed in an inverted-L fashion has become the gold standard for stabilizing a bilateral sagittal split advancement. Various problems emerged, however, showing that the stability necessary for the stabilization of an osteotomy site cannot be directly compared with that of a fracture. Other problems encountered were difficulties in positioning the fragments in new sites, which resulted in malposition of the condyle. This led to the term 'immediate postoperative relapse'. In addition, pain and dysfunction of the temporomandibular joint (TMJ) complicated the treatment and made the target of long-term stability difficult to achieve.

In this current study a comparison between 3 positional screws in comparison with the adjustable plate in conjunction with 2 positional screws will be used in a group of patients suffering from retrognathia and will be treated by BSSRO, thus the investigators are using the advantage of the inherent adjustability of the plate intraoperatively with the good fixation and the stability inherent in the bicortical screws short term stability. This will be evaluated both clinically and cephalometrically.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from mandibular retrognathia (anteroposterior deficient mandible)
* Patients should be free from any systemic disease that may affect normal healing, and predictable outcome

Exclusion Criteria:

* Patients with any systemic disease that may affect normal healing
* Intra-bony lesions or infections that may retard the osteotomy healing
* Uncooperative Patient with bad oral hygiene

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
cephalometric analysis to measure angles(degrees) | (an xray preoperative, immediate postoperative, 6 weeks and 6 months)
cephalometric analysis to measure lines(mm) | (an xray preoperative, immediate postoperative, 6 weeks and 6 months)

SECONDARY OUTCOMES:
operation time in minutes | intraoperative timing during surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Sickels JE, Peterson GP, Holms S, Haug RH. An in vitro comparison of an adjustable bone fixation system. J Oral Maxillofac Surg. 2005 Nov;63(11):1620-5. doi: 10.1016/j.joms.2005.06.008. PMID 16243179
- [Result] Joos U. An adjustable bone fixation system for sagittal split ramus osteotomy: preliminary report. Br J Oral Maxillofac Surg. 1999 Apr;37(2):99-103. doi: 10.1054/bjom.1997.0081. PMID 10371309
- [Result] Peterson GP, Haug RH, Van Sickels J. A biomechanical evaluation of bilateral sagittal ramus osteotomy fixation techniques. J Oral Maxillofac Surg. 2005 Sep;63(9):1317-24. doi: 10.1016/j.joms.2005.05.301. PMID 16122596